CLINICAL TRIAL: NCT04172857
Title: Treatment of Malignant Glaucoma Secondary to Cataract Surgery Combined With Goniosynechialysis by Anterior Vitrectomy From Two Different Approaches
Brief Title: Treatment of Malignant Glaucoma by Anterior Vitrectomy From Two Different Approaches
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, Researcher；clinical research center, Wenzhou Medical University
Other Study IDs: QZB-MG
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Glaucoma Secondary
MeSH Terms: interventions — Iridectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: anterior vitrectomy combined with hyaloidotomy, zonulectomy and iridectomy — First, a 23-G incision was made at the peripheral inferior temporal sector of the cornea and connected with an anterior chamber infusion cannula. Another corneal incision was made at the superior temporal sector or superior nasal sector, and Viscoat® (Bausch & Lomb, Shandong, China) was infused though the incision to fill the anterior chamber. Iridotomy was performed through the incision using Wescott scissors and toothed forceps. Hyaloidectomy and zonulectomy were performed through a peripheral iris defect using an anterior chamber approach to set up a pathway between the anterior chamber and the vitreous cavity. We repeatedly carried out vitrectomy around the pathway to reduce the risk of postoperative re-obstruction of the tunnel created.

SUMMARY:
To compare the surgical outcomes of treating phacoemulsification with intraocular lens implantation combined with goniosynechialysis (Phaco-IOL-GSL) associated malignant glaucoma (MG), using different incision sites in anterior vitrectomy combined with hyaloidotomy, zonulectomy, and iridectomy (VHZI).

ELIGIBILITY:
Inclusion Criteria:

* MG was diagnosed based on the presence of a central and peripheral shallow anterior chamber with normal or elevated intraocular pressure (IOP).

Exclusion Criteria:

* The diagnosis was made only after confirming the absence of choroidal detachment or hemorrhage and posterior segment mass lesion, using B-scan ultrasonography or ophthalmoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The medical records of all patients who developed clinical evidence of MG after Phaco-IOL-GSL, at the Affiliated Eye Hospital of Wenzhou Medical University from May 2015 to February 2018, were reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Relapse of MG | follow up: 3 to 31 months
  MG relapse after the anterior vitrectomy combined with hyaloidotomy, zonulectomy, and iridectomy (VHZI).

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Qian Z, Chan YK, Wei L, Zheng B, Nie L, Pan W. Evaluation of Two Different Anterior Vitrectomies for Fluid Misdirection Syndrome Secondary to Cataract Surgery Combined with Goniosynechialysis. J Ophthalmol. 2020 Mar 23;2020:1934086. doi: 10.1155/2020/1934086. eCollection 2020. PMID 32280517